CLINICAL TRIAL: NCT07044817
Title: Determining the Compliance With the Guidelines of Physiotherapists' and Physiotherapy Internship Students' Attitudes Regarding the Treatment Approach of Post-Stroke Patients
Brief Title: Adherence to Stroke Rehabilitation Guidelines Among Physical Therapists and Internship Students
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ibrahim Magdy Ibrahim Ibrahim Elboraey, Principal Investigator, Medipol University
Other Study IDs: E-10840098-202.3.02-2920
Record Dates: First submitted 2025-05-30; First posted 2025-07-01 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Evidence Based Practice; Stroke; Physical Therapist
Keywords: Stroke Rehabilitation; Evidence Based Practice; Clinical Practice Guidelines; Physical Therapists; Internship and Residency; Professional Practice Gaps; Health Knowledge; Attitudes; Practice; Turkey; Cross Sectional Studies; Treatment Adherence and Compliance; Health Services Accessibility; Physical Therapy Modalities; Clinical Competence; Practice Guidelines; Physical Therapy
MeSH Terms: conditions — Stroke; Behavior; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Licensed Physiotherapists: This group includes licensed physiotherapists in Turkey with at least one year of clinical experience treating post-stroke patients. Participants will complete a survey assessing their adherence to clinical practice guidelines, attitudes toward evidence-based practice, and perceived barriers in stroke rehabilitation.
  Interventions: Behavioral: Stroke Rehabilitation Guideline Adherence Survey
- Physiotherapy Internship Students: This group includes final-year physiotherapy students currently completing their clinical internships in Turkey. Participants will complete a survey evaluating their knowledge, attitudes, and challenges related to stroke rehabilitation and the use of evidence-based guidelines.
  Interventions: Behavioral: Stroke Rehabilitation Guideline Adherence Survey

INTERVENTIONS:
Behavioral: Stroke Rehabilitation Guideline Adherence Survey — This intervention consists of a structured online survey, the Stroke Rehabilitation Guideline Adherence Survey, designed to assess physiotherapists' and physiotherapy internship students' adherence to stroke rehabilitation clinical practice guidelines, their attitudes toward implementing evidence-based post-stroke care, and the perceived barriers-such as time constraints, limited resources, or insufficient training-that influence their compliance. No clinical treatments or procedures are administered; the sole "intervention" is the delivery of this comprehensive questionnaire.

SUMMARY:
The goal of this observational study is to learn about adherence to the 2024 VA/DoD Clinical Practice Guidelines for Stroke Rehabilitation among Turkish physiotherapists and internship students treating post-stroke patients. The main questions it aims to answer are:

1. What is the level of adherence to these evidence-based stroke rehabilitation guidelines?
2. How does guideline adherence differ between licensed physiotherapists and internship students?
3. What are the most significant barriers to using these guidelines (e.g., lack of time or resources)?

Researchers will compare responses from:

* Licensed physiotherapists** (with ≥1 year of experience)
* 4th-year physiotherapy students** (during internships) to understand differences in compliance.

Participants will:

* Complete an online survey about their:
* Use of guideline-recommended interventions (e.g., task-specific training, technology).
* Attitudes toward evidence-based practice.
* Perceived barriers to applying the guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Licensed physiotherapists with ≥1 year of clinical experience.
* 4th-year physiotherapy students enrolled in accredited Turkish universities.

Exclusion Criteria:

* Incomplete survey responses (<80% completion).
* Participants outside Turkey.
* Licensed therapists working in non-clinical roles (e.g., administrative, research-only).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Licensed physical therapists and final-year physiotherapy internship students from diverse clinical and academic settings across Turkey will be recruited via email invitations, academic program coordinators, and online professional forums such as WhatsApp and LinkedIn, ensuring a representative community-based sample of practitioners and trainees involved in post-stroke care.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Guideline Adherence Between Licensed Physical Therapists and Internship Students | At the time of survey completion (Baseline)
  Analysis of differences in adherence scores between licensed physical therapists and internship students to identify any significant variation in guideline implementation practices.

SECONDARY OUTCOMES:
Adherence to Stroke Rehabilitation Guidelines Among Licensed Physical Therapists and Internship Students | At the time of survey completion (Baseline)
  Assessment of the level of adherence to evidence-based stroke rehabilitation guidelines among licensed physical therapists and 4th-year internship students. This is measured by responses to a structured questionnaire evaluating compliance with specific clinical practice recommendations.
Identification of Barriers to Implementing Evidence-Based Stroke Rehabilitation Guidelines | At the time of survey completion (Baseline)
  Evaluation of the challenges and barriers reported by physical therapists and internship students in applying evidence-based stroke rehabilitation guidelines and advanced techniques, as collected through the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen Şahin, Dr. Assistant Professor, Study Director — Department of Physiotherapy and Rehabilitation/Istanbul Medipol University
Locations (1):
- Medipol University, Istanbul, Beykoz/İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cormican A, Hirani SP, McKeown E. Healthcare professionals' perceived barriers and facilitators of implementing clinical practice guidelines for stroke rehabilitation: A systematic review. Clin Rehabil. 2023 May;37(5):701-712. doi: 10.1177/02692155221141036. Epub 2022 Dec 7. PMID 36475911
- [Background] Iles R, Davidson M. Evidence based practice: a survey of physiotherapists' current practice. Physiother Res Int. 2006 Jun;11(2):93-103. doi: 10.1002/pri.328. PMID 16808090
- [Background] Jette DU, Bacon K, Batty C, Carlson M, Ferland A, Hemingway RD, Hill JC, Ogilvie L, Volk D. Evidence-based practice: beliefs, attitudes, knowledge, and behaviors of physical therapists. Phys Ther. 2003 Sep;83(9):786-805. PMID 12940766
- [Background] Korner-Bitensky N, Desrosiers J, Rochette A. A national survey of occupational therapists' practices related to participation post-stroke. J Rehabil Med. 2008 Apr;40(4):291-7. doi: 10.2340/16501977-0167. PMID 18382825
- [Background] Rochette A, Korner-Bitensky N, Desrosiers J. Actual vs best practice for families post-stroke according to three rehabilitation disciplines. J Rehabil Med. 2007 Sep;39(7):513-9. doi: 10.2340/16501977-0082. PMID 17724549
- [Background] Dumoulin C, Korner-Bitensky N, Tannenbaum C. Urinary incontinence after stroke: identification, assessment, and intervention by rehabilitation professionals in Canada. Stroke. 2007 Oct;38(10):2745-51. doi: 10.1161/STROKEAHA.107.486035. Epub 2007 Sep 6. PMID 17823380
- [Background] Paci M, Faedda G, Ugolini A, Pellicciari L. Barriers to evidence-based practice implementation in physiotherapy: a systematic review and meta-analysis. Int J Qual Health Care. 2021 Jun 26;33(2):mzab093. doi: 10.1093/intqhc/mzab093. PMID 34110410
- [Background] Salbach NM, Guilcher SJ, Jaglal SB, Davis DA. Determinants of research use in clinical decision making among physical therapists providing services post-stroke: a cross-sectional study. Implement Sci. 2010 Oct 14;5:77. doi: 10.1186/1748-5908-5-77. PMID 20946678
- [Background] Gale BV, Schaffer MA. Organizational readiness for evidence-based practice. J Nurs Adm. 2009 Feb;39(2):91-7. doi: 10.1097/NNA.0b013e318195a48d. PMID 19190426
- [Background] Sackett DL, Rosenberg WM, Gray JA, Haynes RB, Richardson WS. Evidence based medicine: what it is and what it isn't. BMJ. 1996 Jan 13;312(7023):71-2. doi: 10.1136/bmj.312.7023.71. No abstract available. PMID 8555924
- [Background] Donkor ES. Stroke in the 21st Century: A Snapshot of the Burden, Epidemiology, and Quality of Life. Stroke Res Treat. 2018 Nov 27;2018:3238165. doi: 10.1155/2018/3238165. eCollection 2018. PMID 30598741
- See also: This website provides clinical practice guidelines on stroke rehabilitation published by the Veterans Affairs/Department of Defense (VA/DoD). It offers evidence-based recommendations relevant to the study protocol on post-stroke rehabilitation adherence — https://www.healthquality.va.gov/guidelines/rehab/stroke/